CLINICAL TRIAL: NCT07272525
Title: Research Study for Single-Patient Treatment of Cree Leukoencephalopathy/Vanishing White Matter Disease
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Genevieve Bernard, MD, MSc, FRCPc, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-10780 (CLE-ABBV-CLS-7262)
Record Dates: First submitted 2024-10-11; First posted 2025-12-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cree Leukoencephalopathy; Vanishing White Matter
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- N=1 trial (Experimental): N=1 trial
  Interventions: Drug: Fosigotifator (FGT/ABBV-CLS-7262)

INTERVENTIONS:
Drug: Fosigotifator (FGT/ABBV-CLS-7262) — This study aims to provide under compassionate use program access to an investigational drug (FGT) for a patient diagnosed with Cree Leukoencephalopathy (CLE)/Vanishing White Matter (VWM) which has no treatment options currently available. The study will also evaluate the risk/benefit of FGT in slowing or halting the progression of white matter degeneration in a patient with CLE. By targeting the underlying pathophysiological mechanisms of white matter damage, FGT is expected to alleviate neurological symptoms and improve the quality of life for the patient. The outcomes of this study could provide critical insights into the disease's management and pave the way for the development of targeted therapies, ultimately offering hope to a population with limited treatment options.

SUMMARY:
Cree Leukoencephalopathy (CLE) is a rare and fatal neurodegenerative disorder predominantly affecting the Cree population in Northern Quebec. Characterized by progressive white matter degeneration, this condition leads to severe neurological impairment and decline, leading to premature death. Despite its significant impact on the affected population, there are currently no effective treatments for CLE. CLE is caused by a single founder pathogenic variant in the EIF2B5 gene and is therefore allelic to VWM.

Fosigotifator (FGT, ABBV-CLS-7262) has been developed and its safety and efficacy are currently being studied in a multi-center Phase 1b/2 clinical trial for Vanishing White Matter (VWM) by Calico in collaboration with AbbVie.

This study aims to provide under compassionate use program access to an investigational drug (FGT) for a patient diagnosed with CLE/VWM disease which has no treatment options currently available. The study will also evaluate the risk/benefit of FGT in slowing or halting the progression of white matter degeneration in a patient with CLE. By targeting the underlying pathophysiological mechanisms of white matter damage, FGT is expected to alleviate neurological symptoms and improve the quality of life for the patient. The outcomes of this study could provide critical insights into the disease's management and pave the way for the development of targeted therapies, ultimately offering hope to a population with limited treatment options.

ELIGIBILITY:
Inclusion Criteria:

The patient meets the following criteria:

* Molecularly confirmed diagnosis of CLE
* Pre-symptomatic or early symptomatic patient
* Signed informed consent from the Legal Guardians/caregivers (parents)

Exclusion Criteria:

N/A

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient survival or need for continuous ventilatory support at 2 years | 3 years
  Patient survival (yes/no) or need for continuous ventilatory support (yes/no) at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided